CLINICAL TRIAL: NCT03141749
Title: Incidence and Predictors of Venous Thromboembolism in Myotonic Dystrophy
Brief Title: Venous Thromboembolism in DM1
Acronym: DM1-VTE
Status: Completed | Type: Observational
Sponsor: Institut de Myologie, France (Other)
Responsible Party: Sponsor
Other Study IDs: Institutmyologie
Record Dates: First submitted 2017-05-03; First posted 2017-05-05 (Actual); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Venous Thromboembolism; Pulmonary Embolism; Deep Vein Thrombosis; Myopathy; Myotonic Dystrophy 1
MeSH Terms: conditions — Venous Thromboembolism; Pulmonary Embolism; Venous Thrombosis; Muscular Diseases; Myotonic Dystrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The risk for venous thromboembolism (VTE) in DM1 and in other inherited myopathies, which can lead to chronic immobilization, are unknown. The purpose of this study is to evaluate incidence of VTE in cohort of patients presenting with DM1 with a comparison to a group of other inheritable myopathies and to a community-based population.

DETAILED DESCRIPTION:
A cohort of more that 2,800 adult patients admitted to our Institutions between January 2000 and November 2014 with genetically proven myopathy will be retrospectively included.

Any information relative to their demographic and genetic characteristics, their muscular functional status and the occurrence of VTE will be collected.

Statistical analysis will be performed to estimate the incidence of venous thromboembolism in this population, to identify predictors of VTE, and to compare its incidence to a community-based population.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Genetically proven myopathy
* Admission in our institutions from January 2000 to November 2014

Exclusion Criteria:

* Patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with genetically proven myopathy
Sampling Method: Non-Probability Sample
Enrollment: 2810 (Actual)
Dates: Start 2000-01 (Actual); Primary Completion 2014-11 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Any episode of pulmonary embolism and/or deep vein thrombosis, diagnosed according to 2011 AHA guidelines on venous thromboembolism management | 14 years

CONTACTS AND LOCATIONS:
Overall Officials: Karim Wahbi, MD, PhD, Principal Investigator — Institut de Myologie, Paris, FRANCE

IPD SHARING:
Plan to Share IPD: Undecided